CLINICAL TRIAL: NCT00788034
Title: A Double-blind, Randomised, Placebo-controlled, Multicentre, Relapse-prevention Study With Lu AA21004 in Patients With Generalized Anxiety Disorder
Brief Title: Relapse-prevention Study With Lu AA21004 (Vortioxetine) in Patients With Generalized Anxiety Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12473A; 2008-001673-15 (EudraCT Number)
Record Dates: First submitted 2008-11-07; First posted 2008-11-10 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2012-12

CONDITIONS: Generalized Anxiety Disorder
Keywords: Relapse prevention; GAD; Maintenance; Double-blind; Multicentre
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — Vortioxetine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lu AA21004 (Experimental)
  Interventions: Drug: Lu AA21004
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lu AA21004 — 5 or 10 mg/day
  Other Names: Vortioxetine
  Arms: Lu AA21004
Drug: Placebo — Once daily
  Arms: Placebo

SUMMARY:
The study will evaluate the long-term maintenance of efficacy of Lu AA21004 in patients with Generalized Anxiety Disorder (GAD) who responded to acute treatment with Lu AA21004.

DETAILED DESCRIPTION:
GAD is a common and disabling mental disorder associated with substantial medical and psychiatric comorbidity and occupational impairment. It is characterized by inappropriate or excessive anxiety and worrying that persists over time for more than six months. Common features include apprehension, with worries about future misfortune; inner tension and difficulty in concentrating; motor tension, with restlessness, tremor and headache; and autonomic anxiety symptoms, with excessive perspiration, dry mouth and epigastric discomfort. GAD is typically a chronic disorder with a high relapse rate and therefore requires effective long-term treatment. Long-term studies are necessary to demonstrate that the short-term effect is maintained.

ELIGIBILITY:
Inclusion Criteria:

The patient has GAD as the primary diagnosis according to DSM-IV-TR criteria (classification code 300.02).

* The patient has a HAM-A total score >=20 at screening and baseline visits
* The patient has a HAM-A score >=2 on both Item 1 (anxious mood) and Item 2 (tension) at screening and baseline visits
* The patient has a MADRS total score <=16 at screening and baseline visits

Exclusion Criteria:

* Any current psychiatric disorder other than GAD as defined in the DSM-IV-TR (assessed with the MINI)
* Any substance disorder (except nicotine and caffeine) within the previous 6 months as defined in the DSM-IV-TR
* Women of childbearing potential not using effective contraception

Other protocol-defined inclusion and exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 459 (Actual)
Dates: Start 2008-10; Primary Completion 2010-06 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Time to relapse | At least 24 weeks

SECONDARY OUTCOMES:
Relapse rates, Hamilton Anxiety Rating Scale (HAM-A), Clinical Global Impression Scale (CGI), MOS SF-36, Sheehan Disability Scale (SDS), Adverse events, Clinical laboratory tests, Vital signs, ECG | At least 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (81):
- Argentina (11):
  - AR010, Buenos Aires
  - AR012, Buenos Aires
  - AR002, Buenos Aires
  - AR008, Buenos Aires
  - AR003, Buenos Aires
  - AR013, Buenos Aires
  - AR004, Córdoba
  - AR015, La Plata
  - AR006, Mendoza
  - AR009, Mendoza
  - AR001, Santa Fé
- Chile (8):
  - CL004, Antofagasta
  - CL001, Coquimbo
  - CL002, Santiago
  - CL003, Santiago
  - CL005, Santiago
  - CL007, Santiago
  - CL008, Santiago
  - CL006, Viña del Mar
- Colombia (7):
  - CO003, Barranquilla
  - CO001, Bogotá
  - CO005, Bogotá
  - CO006, Envigado
  - CO002, Medellín
  - CO007, Medellín
  - CO004, Pareira
- Costa Rica (4):
  - CR002, Escazú
  - CR004, Guadalupe
  - CR001, San José
  - CR003, San Pedro
- Estonia (3):
  - EE001, Tallinn
  - EE004, Tallinn
  - EE002, Tartu
- Finland (12):
  - FI006, Espoo
  - FI008, Helsinki
  - FI001, Helsinki
  - FI004, Helsinki
  - FI011, Helsinki
  - FI010, Helsinki
  - FI005, Juväskylä
  - FI012, Kuopio
  - FI002, Oulu
  - FI009, Rauma
  - FI003, Turku
  - FI007, Turku
- France (11):
  - FR011, Arcachon
  - FR010, Caen
  - FR016, Douai
  - FR012, Nantes
  - FR004, Nîmes
  - FR013, Palaiseau
  - FR007, Rennes
  - FR001, Saint-André-de-Cubzac
  - FR002, Strasbourg
  - FR015, Toulouse
  - FR005, Toulouse
- Hungary (6):
  - HU005, Budapest
  - HU004, Budapest
  - HU002, Budapest
  - HU001, Gyula
  - HU006, Nagykálló
  - HU008, Sopron
- Peru (2):
  - PE003, Lima
  - PE002, Lima
- Russia (5):
  - RU004, Chita
  - RU006, Saint Petersburg
  - RU002, Saint Petersburg
  - RU003, Saint Petersburg
  - RU001, Tomsk
- South Africa (12):
  - ZA006, Bloemfontein
  - ZA004, Cape Town
  - ZA011, Cape Town
  - ZA012, Cape Town
  - ZA003, Cape Town
  - ZA010, Cape Town
  - ZA007, Gauteng
  - ZA001, Gauteng
  - ZA009, Gauteng
  - ZA002, Kempton Park
  - ZA008, KwaZulu Natal
  - ZA005, Welkom

REFERENCES:
- [Result] Baldwin DS, Loft H, Florea I. Lu AA21004, a multimodal psychotropic agent, in the prevention of relapse in adult patients with generalized anxiety disorder. Int Clin Psychopharmacol. 2012 Jul;27(4):197-207. doi: 10.1097/YIC.0b013e3283530ad7. PMID 22475889
- [Derived] Christensen MC, Loft H, Florea I, McIntyre RS. Efficacy of vortioxetine in working patients with generalized anxiety disorder. CNS Spectr. 2019 Apr;24(2):249-257. doi: 10.1017/S1092852917000761. Epub 2017 Oct 30. PMID 29081307